CLINICAL TRIAL: NCT06661148
Title: A Phase 1, Open-Label, 2-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of EPI-003 in Select Nucleos(t)Ide Analogue-Treated, Chronic Hepatitis B Patients.
Brief Title: Study of EPI-003 in Select Nucleos(t)Ide Analogue-Treated, Chronic Hepatitis B Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Epigenic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPI-003-001
Record Dates: First submitted 2024-10-21; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Chronic Hepatitis B; HBV (Hepatitis B Virus)
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EPI-003 group (Experimental): Part A：Single Ascending Dose； Part B：Dose Expansion
  Interventions: Drug: EPI-003

INTERVENTIONS:
Drug: EPI-003 — Intravenous (IV) infusion.

SUMMARY:
This study is an open-label, 2-Part (Single Ascending Dose [Part 1] And Dose Expansion) study that will evaluate the safety of EPI-003 administered to patients with chronic infection with HBV (CHB). EPI-003 is a liver-targeted antiviral therapeutic for intravenous (IV) injection that is capable of precise epigenetic modifications of the HBV genome without causing mutations in the gene sequence itself. This study is designed to determine the safety and pharmacokinetic (PK) and pharmacodynamic (PD) profile of EPI-003 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years (inclusive) at the time of signing the informed consent.
2. Body mass index (BMI) ≥ 18 kg/m2 and ≤ 35 kg/m2 at Screening, and body weight of ≤ 120 kg.
3. Chronic HBV infection for ≥ 6 months prior to Screening (eg, positive for serum HBsAg, HBV DNA, HBeAg for ≥ 6 months ) or serum immunoglobulin M (IgM) anti-HBc (hepatitis B core antibody) negative at Screening; AND Baseline HBsAg positive at Screening.
4. Has received treatment with a NA (entecavir, tenofovir disoproxil fumarate or tenofovir alafenamide) as a stable dose for ≥ 6 months before Screening and plans to continue at the same dose level for the duration of the study. Participants may be on other NAs but require Sponsor approval before enrolment.
5. HBV DNA < LLOQ (according to local guidelines) for ≥ 6 months and at Screening
6. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 × upper limit of normal (ULN) at Screening.
7. Able and willing to attend the necessary visits to the study site.
8. Able and willing to provide written informed consent after the nature of the study has been explained and prior to the commencement of any study procedures.

Exclusion Criteria:

1. Evidence or history of liver disease of non-HBV aetiology.
2. Previous history or current diagnosis of significant liver fibrosis or cirrhosis
3. Liver ultrasound or other imaging with findings suggestive of HCC at any time.
4. Participants with serum alpha-fetoprotein (AFP) ≥ 200 ng/mL at Screening.
5. Positive test result for HIV-1 or HIV-2 that suggests a concurrent infection at Screening.
6. History of acute febrile illness, symptomatic viral, bacterial, or fungal infection within 1 week before Day 1.
7. History of receiving HBV vaccine or other HBV-targeted therapeutic within the 6 months before Day 1.
8. Previous treatment with an HBV-targeted treatment other than NAs within the 6 months before Day 1 or planned use during the study.
9. Any of the laboratory values at Screening (Screening laboratory tests may be repeated once for values thought to be erroneous OR not clinically significant as per the PI):
10. Immunodeficient or autoimmune conditions due to disease.
11. Chronic treatment with immunosuppressants.
12. Any history of unexplained blackouts, fainting episodes, significant arrythmias, clinically significant abnormality of ECG, marked QT abnormalities, or any known risk factors for Torsade de Points
13. History of anaphylaxis, hypersensitivity, or significant drug allergies.
14. Received any antiplatelet or antithrombotic therapy.
15. History of thrombophilia or history of a positive genetic test for Factor V Leiden and/or prothrombin 20210.
16. Known or suspected intolerance or hypersensitivity to the IP components.
17. Have received any other IP within 30 days or 5 half-lives of Day 1.
18. Have received any vaccination within 14 days prior to Day 1 or vaccination planned for 3 months following administration of IP.
19. Received any medications or other treatments that may adversely affect the immune system.
20. Excess alcohol consumption within 3 months of Screening.
21. Significant drug abuse/addiction within 3 months of Screening.
22. Any safety concern or personal condition that is inappropriate for study participation per the Investigator's judgement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | From Baseline through to Day 28 postdose
  Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Change from baseline at different follow-up time points for HBsAg, HBsAb, HBV DNA, HBV pgRNA and HBcrAg | From Baseline (predose on Day 1) at Day 3, Day 7, Day 14, Day 28, Day 56, Day 84, Day 112, and Day 182, and Day 365 postdose for the following parameters
  Change from baseline at different follow-up time points for HBsAg, HBsAb, HBV DNA, HBV pgRNA and HBcrAg
Evaluation of maximum observed concentration (Cmax) | Day 1, Day 3, Day 14, and Day 28
  Evaluation of maximum observed concentration (Cmax)
Evaluation of maximum observed concentration (tmax) | Day 1, Day 3, Day 14, and Day 28
  Evaluation of maximum observed concentration (tmax)
Evaluation of terminal elimination half-life (t1/2) | Day 1, Day 3, Day 14, and Day 28
  Evaluation of terminal elimination half-life (t1/2)

OTHER OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs). | Up to day365
  Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Locations (4):
- Epigenic Therapeutics Investigational Site, Westmead, New South Wales, Australia
- Epigenic Therapeutics Investigational Site, Hong Kong, China
- New Zealand (2):
  - Epigenic Therapeutics Investigational Site, Grafton, Auckland
  - Epigenic Therapeutics Investigational Site, Christchurch

IPD SHARING:
Plan to Share IPD: No